CLINICAL TRIAL: NCT05531786
Title: Phase I/II Study of Pacritinib, A JAK2/IRAK1/CSF1R Inhibitor, in Refractory Chronic Graft-Versus-Host Disease (cGVHD) After Allogeneic Hematopoietic Stem Cell Transplantation (HSCT)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10000643; 000643-C
Record Dates: First submitted 2022-09-03; First posted 2022-09-08 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11-21

CONDITIONS: Graft vs Host Disease
Keywords: Anti-Inflammatory; Fibrosis; Inflammation; Refractory; Systemic Therapy
MeSH Terms: conditions — Graft vs Host Disease; Fibrosis; Inflammation | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 2 - Low-dose (Experimental): Expansion dosing to evaluate the efficacy of pacritinib 100 mg PO BID
  Interventions: Drug: Pacritinib
- Arm 3 - High-dose (Experimental): Expansion dosing to evaluate the efficacy of pacritinib 200 mg PO BID
  Interventions: Drug: Pacritinib
- Escalating doses of treatment (Experimental): Escalating doses of pacritinib to confirm safety in cGVHD
  Interventions: Drug: Pacritinib

INTERVENTIONS:
Drug: Pacritinib — Pacritinib will be given as 100 mg or 200 mg tablets to be taken orally twice daily (12 hours apart) on days 1-28 of a 28 day cycle. Morning and evening should be taken at approximately the same time of day.

SUMMARY:
Background:

Chronic graft-versus-host disease (cGVHD) is an immune system disorder that can occur in people who have had a stem cell transplant. cGVHD can affect multiple organs and increase risk of disability and death. New treatments are needed to treat cGVHD after stem cell transplant.

Objective:

To test a drug (pacritinib) in people with moderate or severe cGVHD that has not responded to previous treatment.

Eligibility:

People aged 18 years and older with moderate or severe cGVHD that has not responded to 2 or more lines of previous treatment.

Design:

Participants will be screened. They will have blood and urine tests. They will have tests of their heart and lung function. They may also have a CT scan. Some may have other specialized tests.

Participants will take the study drug at home every day. Pacritinib is a capsule taken by mouth. The study doctor will determine the dosage and schedule.

Participants will keep a medication diary. They will record the date and time of each drug dose and any missed doses.

Participants will visit the clinic every 2 weeks for the first 4 months. Then they will visit the clinic once every 4 weeks. They will have blood and urine tests. During some visits, other screening tests will be repeated, and participants will fill out questionnaires about their quality of life. Photographs may be taken of skin rashes and joints affected by cGVHD.

Participants will give saliva samples. Optional biopsies may be taken of the skin and mouth.

Participants will take pacritinib for 6 to 12 months if no side effects develop. Follow-up visits will continue for up to 2 years.

...

DETAILED DESCRIPTION:
Background:

* Chronic GVHD (cGVHD) is a multi-organ disorder characterized by immune dysregulation, impaired organ function, and decreased survival for hematopoietic stem cell transplantation (HSCT) patients.
* The JAK-STAT pathway plays an important role in immune cell development and function, including antigen presenting cells, B- and T-cells, and its activation leads to a cascade promoting a proinflammatory cytokine milieu.
* Pacritinib is a JAK2/IRAK1/CSF1R/FLT3 inhibitor, with an established safety and efficacy profile in the treatment of myeloproliferative neoplasms (myelofibrosis) and of acute GVHD.
* Pacritinib s immunomodulatory effects suggest therapeutic benefit for cGVHD, without abrogating the graft-versus-leukemia effect after HSCT.

Objectives:

* Phase I: to determine the safety of pacritinib in participants with refractory cGVHD
* Phase II: to determine the efficacy of pacritinib in participants with refractory cGVHD

Eligibility:

* Moderate or severe cGVHD (after allogeneic hematopoietic stem cell transplantation) diagnosed and staged per NIH criteria.
* cGVHD that did not respond to at least two prior lines of systemic therapy.
* Age >=18 years.
* If participant is taking systemic therapy for cGVHD at the time of enrollment, they must be on stable or tapering doses in the preceding 4 weeks.
* Participants must have adequate organ and marrow function.

Design:

* This Phase I/II study will use a modified 3+3 dose-escalation design, with two planned dose levels of pacritinib, followed by a small efficacy evaluation in a randomized phase II design.
* Pacritinib will be given taken orally once or twice daily (based on dose level) on days 1- 28 of a 28-day cycle.
* Pacritinib treatment will continue for up to 12 months. cGVHD response will be evaluated at 6 weeks, and 3, 6, 9 and 12 months from the start of pacritinib. All participants will be followed through 2 years post-initiation of pacritinib.
* The accrual ceiling set at 50 participants.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Moderate or severe cGVHD (after allogeneic hematopoietic stem cell transplantation) diagnosed and staged per NIH criteria
2. cGVHD that did not respond to >=2 lines of prior systemic therapy.

   Disease that has failed prior systemic therapy will be defined as follows:

   a) For prior corticosteroid-containing regimens, disease that:

   i) recurs after achievement of a CR, or

   ii) progresses after achievement of a PR, or

   iii) progresses after at least 1 week of prednisone equivalent of 1 mg/kg/day, or

   iv) is stable and persistent after at least 4 weeks of a prednisone equivalent of 0.5 mg/kg/day

   OR,

   b) For other systemic therapies, disease that:

   i) recurs after achievement of CR, or

   ii) progresses after achievement of a PR, or

   iii) is stable and persistent despite 4 weeks of therapeutic dosing of systemic therapy
3. Karnofsky performance score >=60%
4. Age >=18 years.
5. If participant is taking systemic therapy for cGVHD at the time of enrollment, they must be on a stable or tapering dose in the preceding 4 weeks.
6. Participants must have adequate organ and marrow function as defined below:

   * absolute neutrophil count >=1,000/mcL
   * platelets >=50,000/mcL
   * total bilirubin <=1.5 X institutional upper limit of normal

   OR

   <=3 X institutional upper limit of normal in participants with Gilbert's syndrome
   * AST(SGOT)/ALT(SGPT) <=3 X institutional upper limit of normal
   * creatinine clearance >=50 mL/min/1.73 m^2 per Cockroft-Gault
7. Primary malignancy for which the participant received transplant has been in complete clinical remission and stable for 3 months prior to enrollment on study.
8. Individuals of child-bearing potential (IOCBP) and individuals able to father a child with a partner able to become pregnant who are sexually active must agree to use one (1) highly effective (e.g., intrauterine device [IUD], surgical) or two (2) effective forms of contraception (e.g., barrier method) at study entry, for the duration of study treatment, and for at least 90 days after last study drug exposure.
9. Ability of participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

1. Acute GVHD that is active as defined by exhibiting current signs or symptoms of disease without any chronic GVHD (classic and late-acute GVHD per NIH consensus criteria); participants with a clinical presentation consistent with overlapping acute GVHD with concurrent chronic GVHD will be eligible
2. Treatment with ruxolitinib, or ibrutinib within the for <= 14 days prior to treatment initiation.
3. Active HIV-1 (detectable HIV viral load), or Hepatitis B (HBV) and/or Hepatitis C (HCV) infection (positive HBV or HCV viral load in the setting of positive HBV core antibody or surface antibody or HCV antibody).
4. Participants with the following cardiac conditions at screening:

   * symptomatic congestive heart failure
   * unstable angina pectoris
   * uncontrolled cardiac dysrhythmias
   * QTc(F) prolongation >450 ms or other factors that increase the risk for QT prolongation (i.e., heart failure, or a history of long QT interval syndrome).
5. Left ventricular ejection fraction <= 50% by transthoracic echocardiogram (TTE) at screening.
6. Participants with poor pulmonary function as defined by a forced expiratory volume in the first second (FEV1) <= 39% calculated using the USA-ITS-NIH equation.
7. Participants with evidence of ongoing hemorrhage, active signs/symptoms of bleeding, or history of severe bleeding complications in the one year prior to enrollment.
8. Concurrent treatment with any other investigational agents.
9. Concurrent use of strong CYP3A4 inducers or inhibitors, must stop 2 weeks prior study drug initiation.
10. Known hypersensitivity to JAK inhibitors.
11. Participants who are unwilling to accept blood transfusions.
12. Pregnancy or breastfeeding.
13. Participants with any active, uncontrolled viral, bacterial, or fungal infection are excluded.
14. Other malignancy except non-melanoma skin cancer or carcinoma in situ of the cervix or breast which requires active treatment.
15. Uncontrolled intercurrent illness evaluated by history, physical exam and chemistries or situation that would limit compliance with study requirements.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2027-07-22 (Estimated); Study Completion 2027-07-22 (Estimated)

PRIMARY OUTCOMES:
Phase I: Safety of pacritinib in refractory cGVHD. | 60 days
  grades and types of toxicity reported at each dose level. The overall estimate of the fraction of patients who have a DLT at the MTD will be reported.
Phase II: Overall response rate (ORR) | 6 months
  the fraction with clinical responses reported separately by arm, with a separate 95% confidence interval for each cohort.

SECONDARY OUTCOMES:
Phase I: Pharmacokinetics (PK) | every 3 months through up to 12 months of treatment
  The secondary endpoint for PK properties includes measures such as AUC, half-life, and steady-state concentration.
Phase 2: Safety | every 3 months through up to 12 months of treatment
  Toxicities identified from day 1 of study drug, collected every 2 weeks through cycle 4, then per cycle through 30 days after the study drug administration. AEs are reported by type and grade
Phase 2: Clinical outcomes | every 3 months through up to 12 months of treatment
  Rate of reduction and/or discontinuation of immunosuppressive therapy; response by organ system; time to response; duration of best response; and, failure-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Najla El Jurdi, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@@@@@@@ All collected IPD will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000643-C.html